CLINICAL TRIAL: NCT01060332
Title: The Body Constitution and Quality of Life of Diabetic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Chia-I Tsai/Visiting Staff, Traditional Chinese Medicine Department
Other Study IDs: grb03484888
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- diabetics
  Interventions: Other: Body Constitution Questionnaire

INTERVENTIONS:
Other: Body Constitution Questionnaire — Body Constitution Questionnaire was a tool for the study of objective evaluation of diagnostics of Traditional Chinese Medicine. It has been well developed with good validation and consistency.
  Other Names: BCQ

SUMMARY:
Diabetic Mellitus is the fifth cause of death by the report of Department of Health in 2008, and it often cause the severity of other chronic diseases. Neuropathy, retinopathy and renopathy are the most prevalent complications of DM, and they often influence the quality of life.

300 patients with Diabetic neuropathy will be recruited in Taichung Veterans General Hospital endocrine and metabolism clinics. Body Constitution Questionnaire(BCQ), Diabetes Impact Measurement Scales(DIMS), Short Form -36(SF-36) will be asked to filled up, neurological examination (NE), AC sugar, HbA1c, lipid profiles, liver and kidney functions will be measured in order to evaluate the correlation between body constitution and quality of life on patients with diabetic complication.

DETAILED DESCRIPTION:
Diabetic Mellitus is the fifth cause of death by the report of Department of Health in 2008, and it often cause the severity of other chronic diseases. Neuropathy, retinopathy and renopathy are the most prevalent complications of DM, and they often influence the quality of life.

Traditional Chinese Medicine was often prescribed to treat diabetic complications and improve the quality of life .But the study of objective evaluation of diagnostics of Traditional Chinese Medicine was few . It is important to analyze population of specific disease with well developed Traditional Chinese Medicine diagnostic tool with good validation and consistency.

300 patients with Diabetic neuropathy will be recruited in Taichung Veterans General Hospital endocrine and metabolism clinics. Body Constitution Questionnaire(BCQ), Diabetes Impact Measurement Scales(DIMS), Short Form -36(SF-36) will be asked to filled up, neurological examination (NE), AC sugar, HbA1c, lipid profiles, liver and kidney functions will be measured in order to evaluate the correlation between body constitution and quality of life on patients with diabetic complication.

ELIGIBILITY:
Inclusion Criteria:

* There is a history of diabetes and the injection or taking hypoglycemic agents.
* Aged 20 years of age, not limit to male or female .
* Consciousness clear, subjects are willing to sign consent after stating research purpose and process.

Exclusion Criteria:

* Took the Chinese medicine within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health Center for Diabetic Patient
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Body Constitution Questionnaire, BCQ | 1 month

SECONDARY OUTCOMES:
Diabetes Impact Measurement Scales | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jia-I Tsai, master, Principal Investigator — Traditional Chinese Medicine
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan